CLINICAL TRIAL: NCT01350882
Title: Phase III Study of Impact of Treatment With Rituximab on the Progression of Humoral Acute Rejection After Renal Transplantation
Brief Title: Impact of Treatment With Rituximab on the Progression of Humoral Acute Rejection After Renal Transplantation
Acronym: RITUX-ERAH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PHRN07-YL RITUXERAH
Record Dates: First submitted 2010-02-04; First posted 2011-05-10 (Estimated); Last update posted 2025-12-26 (Actual); Status verified 2018-02

CONDITIONS: Humoral Rejection in Kidney Transplantation
Keywords: kidney transplantation; acute humoral rejection; rituximab
MeSH Terms: interventions — Rituximab; Sodium Citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Patients randomized into the arm blind A. Rituximab is allowed as additional treatment from J12, within the limit of 2 infusions of rituximab. In case of insufficient efficacy of the treatment of acute humoral rejection, investigators may propose an additional infusion of rituximab from J12, without patient withdrawn. In this case (2nd infusion effective in group A and 1st infusion effective group B), a additional consultation (CS) will be provided as part of the study 7 days after infusion. In case of insufficient efficacy of the treatment,in fairness to care for patients between the 2 treatment groups, the investigators may propose to a 3rd infusion patients in group B (2nd infusion effective for this group). To prevent patients from group A will receive a 3rd infusion of rituximab, unblinding will be applied in this case by the investigator before the administration of additional treatment with rituximab.
  Interventions: Drug: MabThera
- B (Placebo Comparator): Patients randomized into the arm blind B. Rituximab is allowed as additional treatment from J12, within the limit of 2 infusions of rituximab. In case of insufficient efficacy of the treatment of acute humoral rejection, investigators may propose an additional infusion of rituximab from J12, without patient withdrawn. In this case (2nd infusion effective in group A and 1st infusion effective group B), a additional consultation (CS) will be provided as part of the study 7 days after infusion. In case of insufficient efficacy of the treatment,in fairness to care for patients between the 2 treatment groups, the investigators may propose to a 3rd infusion patients in group B (2nd infusion effective for this group). To prevent patients from group A will receive a 3rd infusion of rituximab, unblinding will be applied in this case by the investigator before the administration of additional treatment with rituximab.
  Interventions: Drug: Physiological serum : sodium chloride, sodium citrate

INTERVENTIONS:
Drug: MabThera — MabThera 500mg/50ml I.V. infusion, single dose : 375 mg/m2
  Other Names: rituximab
  Arms: A
Drug: Physiological serum : sodium chloride, sodium citrate — Solution for I.V. infusion Sodium Chloride (pH 6.5), polysorbate 80, sodium citrate (10.0mg/ml)
  Arms: B

SUMMARY:
Assessing the impact of J12 curative treatment with rituximab (375 mg / m² on J5) based on a composite "TREATMENT FAILURE"

ELIGIBILITY:
Inclusion Criteria:

* Patient adult male or female (age 18 years), kidney transplantation for less than one year (transplant from a living donor or deceased), with acute humoral rejection defined by :
* The deterioration of renal function assessed by serum creatinine increase of more than 20% compared to the best value, OR
* In the first 28 days after transplantation, no significant creatinine decrease, AND
* At least 2 of the 3 following criteria:

  * tissue damage such as (a) acute tubular necrosis, (b) presence of monocytes or granulocytes in the CPT and / or glomeruli and / or capillary thrombosis, (c) intimal arteritis / fibrinoid necrosis
  * C4d level of CPT and / or presence of Ig or complement in lesions of fibrinoid necrosis
  * Presence of HLA antibodies directed against the donor. Patient having given his written consent to participate in the clinical trial.

Exclusion Criteria:

* Pregnant or lactating
* Women during their reproductive years without effective contraception,
* A patient with multiple organ transplants,
* Patients with clinically active infection by HCV uncontrolled
* Patients with active infection, or suspected of infection by HIV or HBV, and tuberculosis,
* Patients with heart failure class IV (NYHA) cardiac disease or uncontrolled
* Patients for whom vaccination is scheduled,
* Patient with disabilities did not allow an understanding of the requirements of the test
* Patient in safeguarding justice, guardianship or trusteeship,
* Patient with cons-indication to rituximab (known hypersensitivity to any component or murine protein)
* Patient had previously received rituximab within 3 months before inclusion
* Patient participation in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-10; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
"Treatment failure" grouping at J12: - Loss of graft - Whether improving renal function (defined by the absence of a decrease in creatinine of at least 30% compared to the maximum serum creatinine reached at the RAH) | one year

CONTACTS AND LOCATIONS:
Overall Officials: Yvon LEBRANCHU, Principal Investigator — University Hospital, Tours
Locations (30):
- France (30):
  - Hospital Henri Mondor, Paris, Créteil
  - Hospital, Grenoble, La Tronche
  - Hospital Bicêtre, Paris, Le Kremlin Bicêtre
  - Hospital Lyon Sud, Lyon, Pierre-Benite
  - Hospital Nord, Saint-Etienne, Saint Priez-en-Jarez
  - Hospital Sud, Amiens
  - Hospital, Angers
  - Hospital Saint-Jacques, Besançon
  - Hospital Pellegrin, Bordeaux
  - Hospital, Brest
  - Hospital, Caen
  - Hospital Gabriel Montpied, Clermont-Ferrand
  - Hospital Bocage, Dijon
  - Hospital Calmette, Lille
  - Hospital Dupuytren, Limoges
  - Hospital Edouard Herriot, Lyon
  - Hospital Conception, Marseille
  - Hospital Lapeyronie, Montpellier
  - Hospital Hôtel Dieu, Nantes
  - Hospital Pasteur, Nice
  - Hospital Saint Louis, Paris
  - Hospital Tenon, Paris
  - Hospital Pitié-Salpêtrière, Paris
  - Hospital Necker, Paris
  - Hospital Milétrie Jean Bernard, Poitiers
  - Hospital Maison Blanche, Reims
  - Hospital, Rennes
  - Hospital Bois-Guillaume, Rouen
  - Hospital Civil, Strasbourg
  - Hospital Bretonneau, Tours

REFERENCES:
- [Result] Sautenet B, Blancho G, Buchler M, Morelon E, Toupance O, Barrou B, Ducloux D, Chatelet V, Moulin B, Freguin C, Hazzan M, Lang P, Legendre C, Merville P, Mourad G, Mousson C, Pouteil-Noble C, Purgus R, Rerolle JP, Sayegh J, Westeel PF, Zaoui P, Boivin H, Le Gouge A, Lebranchu Y. One-year Results of the Effects of Rituximab on Acute Antibody-Mediated Rejection in Renal Transplantation: RITUX ERAH, a Multicenter Double-blind Randomized Placebo-controlled Trial. Transplantation. 2016 Feb;100(2):391-9. doi: 10.1097/TP.0000000000000958. PMID 26555944